CLINICAL TRIAL: NCT01412281
Title: Randomized, Parallel-group, Double-blind, Single-center Phase III Study to Assess the Immunogenicity and Safety of the 2011/2012-season Influenza Vaccine Formulated With HA Antigen From Two Suppliers, in Elderly and Young Adult Subjects Using the Current EMA Regulations as Guideline
Brief Title: Immunogenicity and Safety Study to Assess Influenza Vaccine Formulated With Haemagglutinin (HA) Antigen From Two Different Suppliers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ADD-V-A002
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
Keywords: Influenza; Virus; Vaccination; Immunisation
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A - Young adults (Experimental): 1 x 0.5 mL i.m. virosomal influenza vaccine (AdImmune HA Antigen) 2011/2012
  Interventions: Biological: Virosomal influenza vaccine (AdImmune HA Antigen)
- Group B - Young adults (Active Comparator): 1 x 0.5 mL i.m. virosomal influenza vaccine (CSL HA Antigen) 2011/2012
  Interventions: Biological: Virosomal influenza vaccine (CSL HA Antigen)
- Group C - Elderly (Experimental): 1 x 0.5 mL i.m. virosomal influenza vaccine (AdImmune HA Antigen) 2011/2012
  Interventions: Biological: Virosomal influenza vaccine (AdImmune HA Antigen)
- Group D - Elderly (Active Comparator): 1 x 0.5 mL i.m. virosomal influenza vaccine (CSL HA Antigen) 2011/2012
  Interventions: Biological: Virosomal influenza vaccine (CSL HA Antigen)

INTERVENTIONS:
Biological: Virosomal influenza vaccine (AdImmune HA Antigen) — Virosomal influenza vaccine (surface antigen, inactivated, virosome, using AdImmune HA Antigen) 2011/2012, with intramuscular administration, containing per 0.5 mL dose: 15 μg HA antigen of A/California/7/2009 (H1N1)-like virus; 15 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus; 15 μg HA antigen of B/Brisbane/60/2008-like virus
  Arms: Group A - Young adults; Group C - Elderly
Biological: Virosomal influenza vaccine (CSL HA Antigen) — Virosomal influenza vaccine (surface antigen, inactivated, virosome, using CSL HA antigen) 2011/2012 with intramuscular administration, containing per 0.5 mL dose: 15 μg HA antigen of A/California/7/2009 (H1N1)-like virus; 15 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus; 15 μg HA antigen of B/Brisbane/60/2008-like virus
  Arms: Group B - Young adults; Group D - Elderly

SUMMARY:
The purpose of this study is to assess the humoral immune response and safety of the parenteral formulation of the 2010/2011-season virosomal subunit influenza vaccine Inflexal V using two different HA antigen suppliers (AdImmune and CSL), in groups of young and elderly adults, using the EMA (European Medicines Agency) regulation as a guideline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male adults
* Aged ≥18 years on Day 1
* Written informed consent

Exclusion Criteria:

* Acute exacerbation of bronchopulmonary infection (cough, sputum, lung findings) or other acute disease
* Acute febrile illness (≥38.0 °C)
* Prior vaccination with an influenza vaccine (including the H1N1 pandemic swine flu vaccine) in the past 330 days
* Known hypersensitivity to any vaccine component
* Previous history of a serious adverse reaction to influenza vaccine
* History of egg protein allergy or severe atopy
* Known blood coagulation disorder
* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of the study vaccine, incl. oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent (inhaled or topical steroids are allowed)
* Known immunodeficiency (incl. leukemia, cancer, HIV seropositivity)
* Investigational medicinal product received in the past 3 months (90 days)
* Treatment with immunoglobulins or blood transfusion(s) received in the past 3 months (90 days)
* Pregnancy or lactation
* Participation in another clinical trial
* Employee at the investigational site, or spouse and children of the investigator, or relative living in the same household as the investigator and/or are dependent on the investigator
* Suspected non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seiberling, MD, Principal Investigator — Covance Clinical Research Unit AG
Locations (1):
- Covance Clinical Research Unit AG, Allschwil, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 06 October 2011 to 10 November 2011; outpatient study
Period: Overall Study
Arm/Group | ≥18 to ≤60 Years - AdImmune HA Antigen | ≥18 to ≤60 Years - CSL HA Antigen | >60 Years - AdImmune HA Antigen | >60 Years - CSL HA Antigen
Started | 110 | 110 | 110 | 110
Completed | 110 | 110 | 110 | 110
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ≥18 to ≤60 Years - AdImmune HA Antigen | ≥18 to ≤60 Years - CSL HA Antigen | >60 Years - AdImmune HA Antigen | >60 Years - CSL HA Antigen | Total
Number analyzed (Participants) | 110 | 110 | 110 | 110 | 440
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 110 | 110 | 33 | 38 | 291
  >=65 years | 0 | 0 | 77 | 72 | 149
Age Continuous [Mean (Standard Deviation); unit: years] | 39.6 (12.46) | 42.5 (11.98) | 68.4 (5.86) | 67.8 (5.31) | 54.6 (16.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 49 | 48 | 207
  Male | 55 | 55 | 61 | 62 | 233
Region of Enrollment [Number; unit: participants]
  Switzerland | 110 | 110 | 110 | 110 | 440

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer
Description: GMT of HI antibodies and fold-increase in GMT (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters were analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Time Frame: 3 weeks after vaccination (Day 22 ± 2 days)
Population: Intent-to-treat, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: GMT fold increase from baseline
Arm/Group | ≥18 to ≤60 Years - AdImmune HA Antigen | ≥18 to ≤60 Years - CSL HA Antigen | >60 Years - AdImmune HA Antigen | >60 Years - CSL HA Antigen
Number analyzed (Participants) | 110 | 110 | 110 | 110
GMT fold increase from baseline
  GMT fold increase: A/H1N1 | 3.36 [2.78 to 4.07] | 2.61 [2.21 to 3.09] | 2.46 [2.11 to 2.87] | 2.41 [2.04 to 2.85]
  GMT fold increase: A/H3N2 | 2.01 [1.67 to 2.41] | 2.04 [1.76 to 2.36] | 1.65 [1.43 to 1.89] | 1.99 [1.70 to 2.33]
  GMT fold increase: B-strain | 1.75 [1.54 to 1.99] | 1.72 [1.53 to 1.95] | 1.47 [1.33 to 1.62] | 1.32 [1.21 to 1.44]

2. Primary Outcome: Seroprotection
Description: Seroprotection rate, defined as proportion of subjects with HI antibody titer ≥1:40 (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters were analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Time Frame: 3 weeks after vaccination (Day 22 ± 2 days)
Population: Intent-to-treat, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: percentage of seroprotected subjects
Arm/Group | ≥18 to ≤60 Years - AdImmune HA Antigen | ≥18 to ≤60 Years - CSL HA Antigen | >60 Years - AdImmune HA Antigen | >60 Years - CSL HA Antigen
Number analyzed (Participants) | 110 | 110 | 110 | 110
percentage of seroprotected subjects
  Percentage seroprotected subjects: A/H1N1 | 99.1 [95.0 to 100] | 100 [96.7 to 100] | 96.4 [91.0 to 99.0] | 97.3 [92.2 to 99.4]
  Percentage seroprotected subjects: A/H3N2 | 100 [96.7 to 100] | 99.1 [95.0 to 100] | 99.1 [95.0 to 100] | 100 [96.7 to 100]
  Percentage seroprotected subjects: B-strain | 98.2 [93.6 to 99.8] | 100 [96.7 to 100] | 97.3 [92.2 to 99.4] | 95.5 [89.7 to 98.5]

3. Primary Outcome: Seroconversion
Description: Seroconversion rate, defined as proportion of subjects with ≥4-fold increase in HI antibody titer and with a titer of ≥1:40 (The primary endpoints are the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters were analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997)
Time Frame: 3 weeks after vaccination (Day 22 ± 2 days)
Population: Intent-to-treat population, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: percentage of seroconverted subjects
Arm/Group | ≥18 to ≤60 Years - AdImmune HA Antigen | ≥18 to ≤60 Years - CSL HA Antigen | >60 Years - AdImmune HA Antigen | >60 Years - CSL HA Antigen
Number analyzed (Participants) | 110 | 110 | 110 | 110
percentage of seroconverted subjects
  Percentage seroconverted subjects: A/H1N1 | 43.6 [34.2 to 53.4] | 36.4 [27.4 to 46.1] | 23.6 [16.1 to 32.7] | 30.9 [22.4 to 40.4]
  Percentage seroconverted subjects: A/H3N2 | 23.6 [16.1 to 32.7] | 20.0 [13.0 to 28.7] | 16.4 [10.0 to 24.6] | 26.4 [18.4 to 35.6]
  Percentage seroconverted subjects: B-strain | 19.1 [12.2 to 27.7] | 17.3 [10.7 to 25.7] | 8.2 [3.8 to 15.0] | 4.5 [1.5 to 10.3]

4. Secondary Outcome: Number of Participants With Local and Systemic Adverse Events, as a Measure of Safety and Tolerability
Description: Solicited local and systemic AEs, Unsolicited AEs, Tolerability and acceptability
  Unsolicited AEs were collected from baseline (Day 1) to 3 weeks after vaccination (Day 22 ± 2 days).
  Solicited local and systemic AEs were collected by subjects diary from Day 1 (day of vaccination) to Day 4
Time Frame: Baseline (Day 1) and 3 weeks after vaccination (Day 22 ± 2 days)
Population: Safety population, all vaccinated subjects
Measure: Number; unit: participants
Arm/Group | ≥18 to ≤60 Years - AdImmune HA Antigen | ≥18 to ≤60 Years - CSL HA Antigen | >60 Years - AdImmune HA Antigen | >60 Years - CSL HA Antigen
Number analyzed (Participants) | 110 | 110 | 110 | 110
participants
  AEs (unsolicited and unsolicited) | 60 | 52 | 33 | 29
  Unsolicited AEs | 30 | 28 | 17 | 14
  Solicited local AEs | 47 | 32 | 20 | 17
  Solicited systemic AEs | 8 | 10 | 5 | 3

ADVERSE EVENTS:
Arm/Group | ≥18 to ≤60 Years - AdImmune HA Antigen | ≥18 to ≤60 Years - CSL HA Antigen | >60 Years - AdImmune HA Antigen | >60 Years - CSL HA Antigen
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/110 | 0/110 | 1/110
Other Adverse Events (participants affected / at risk) | 60/110 | 52/110 | 33/110 | 29/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ≥18 to ≤60 Years - AdImmune HA Antigen (N=110) | ≥18 to ≤60 Years - CSL HA Antigen (N=110) | >60 Years - AdImmune HA Antigen (N=110) | >60 Years - CSL HA Antigen (N=110)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ≥18 to ≤60 Years - AdImmune HA Antigen (N=110) | ≥18 to ≤60 Years - CSL HA Antigen (N=110) | >60 Years - AdImmune HA Antigen (N=110) | >60 Years - CSL HA Antigen (N=110)
Diarrhoae (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Chills (General disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Erythema (at the injection site) (General disorders) | 11 (11) | 7 (7) | 6 (6) | 9 (9)
Induration (at the injection site) (General disorders) | 6 (6) | 6 (6) | 2 (2) | 4 (4)
Pain (at the injection site) (General disorders) | 44 (44) | 31 (31) | 18 (18) | 12 (12)
Malaise (General disorders) | 6 (6) | 8 (8) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 7 (7) | 2 (2)
Rhinitis (Infections and infestations) | 7 (7) | 5 (5) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 8 (9) | 9 (9) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 90 days from the time submitted to the sponsor for review. The sponsor can make a reasoned request that publication be delayed for up to 3 months from the date of first submission to the sponsor in order to enable the sponsor to protect proprietary information, Intellectual Property, etc.